CLINICAL TRIAL: NCT01079286
Title: Phase I Study of Nelfinavir in Combination With Temsirolimus in the Treatment of Patients With Advanced Cancers, Including Second Line Renal Cell Cancer
Brief Title: Study of Nelfinavir and Temsirolimus in Patients With Advanced Cancers
Acronym: I-NET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Heinz-Josef Klumpen, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMCmedonc09/039
Record Dates: First submitted 2010-02-25; First posted 2010-03-03 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Renal Cell Cancer; Cancer
Keywords: mTOR inhibition; advanced malignancies; pharmacokinetics; Akt inhibition; Advanced malignancies, including metastatic renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Nelfinavir; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nelfinavir and temsirolimus (Experimental): dose escalation
  Interventions: Drug: Nelfinavir and temsirolimus

INTERVENTIONS:
Drug: Nelfinavir and temsirolimus — Nelfinavir tablets of 250mg given twice daily in an escalating dosis schedule, Temsirolimus i.v. given weekly in an escalating dosis schedule
  Other Names: nelfinavir: viracept

SUMMARY:
In the present study the investigators want to explore the safety, pharmacokinetics, and activity of the combination of temsirolimus and nelfinavir, both agents with PI3K /Akt/mTOR inhibiting activity, in patients with advanced malignancies.Temsirolimus has proven anti tumoral activity by mTOR inhibition. Nelfinavir is a potential inhibitor of Akt. Combining both agents might prevent upregulation of the P13k pathway and increase the anti-cancer activity of temsirolimus. The strong CYP3A4 inhibition of nelfinavir and the dependence of temsirolimus on CYP3 A4 metabolism makes a dose finding study essential. The investigators will also look at the prospective value of biomarkers of activity and the outcome of the treatment.

DETAILED DESCRIPTION:
In the past decade, the characterization of human tumours at the molecular level has considerably improved. This has led to the development of targeted therapeutics that inhibit specific molecules and pathways involved in oncogenesis. One of the key pathways that is dysregulated in cancer is the phosphatidylinositol 3'-kinase (PI3K)/Akt/mTOR pathway. This pathway is important for cell growth and survival. In most cancer types this pathway is over-activated leading to proliferation and survival of malignant cells. Inhibition of this pathway is therefore of great therapeutic potential.

Both temsirolimus and nelfinavir are agents with PI3K /Akt/mTOR inhibiting activity. The main active metabolite of temsirolimus is sirolimus that decreases mTOR activity. Inhibition of mTOR activity results in G1 phase cell cycle arrest and subsequent inhibition of tumour growth. Another effect is growth factor downregulation and inhibition of angiogenesis. In addition, mTOR inhibition may exert its anti-tumour effect by inducing apoptosis.

Although inhibitors of mTOR demonstrated clinical activity in tumor types like, mantle cell lymphoma, endometrial carcinoma, and neuro-endocrine tumors, most malignancies are resistant by feedback PI3 kinase activation. Resent data suggest that this tumor escape mechanism can be overcome by dual inhibition of mTOR and PI3 kinase.

Nelfinavir is a well known human immuno-deficiency protease inhibitor with PI3kinase inhibiting activity, via inhibition of Akt, downstream the PI3kinase cascade. Nelfinavir is able to inhibit Akt at concentrations that are achieved in HIV patients at standard antiviral doses. Nelfinavir is therefore a feasable and generally well tolerated agent to be used in combination with temsirolimus to overcome resistance of mTOR inhibition.

Simultaneous inhibition of mTOR/PI3kinase pathway by temsirolimus and nelfinavir is a promising strategy to treat cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological or cytological confirmed malignancies
* ECOG / WHO performance status of 0-2
* Age 18 years
* Life expectancy of at least 3 months
* Minimal acceptable safety laboratory values defined as
* WBC 3.0 x 109 /L
* Platelet count 100 x 109 /L
* Hepatic function as defined by serum bilirubin 1.5 x ULN, ALT or AST 2.5 x ULN, in case of liver metastases 5 x ULN
* Renal function as defined by creatinine < 150μmol/L
* Able and willing to give written informed consent according to ICH/GCP, and national/local regulations.
* Able to swallow and retain oral medication
* Able and willing to undergo blood sampling for pharmacokinetic and pharmacogenetic analysis
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Exclusion Criteria:

* Patients with known alcoholism, drug addiction and/or psychotic disorders in the history that are not suitable for adequate follow up
* Women who are pregnant or breast feeding
* Women of childbearing potential who refuse to use a reliable contraceptive method throughout the study
* Serious concomitant systemic disorder that would compromise the safety of the patient, at the discretion of the investigator
* Any other medical condition that would interfere with study procedures and/or decrease safety of the protocol treatment
* Concomitant use of strong CYP3A4 inhibitors, CYP3A4 inducers or CYP substrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics/pharmacodynamics | During the first 5 weeks of treatment
  PK Nelfinavir: D1, 11, 18, 25, 32 PK Temsirolimus: D4, 11, 18, 25,32
Toxicity profile | Day1 -Day90
  Collection of clinical data according to CTC toxicity criteria

SECONDARY OUTCOMES:
Objective response to treatment | Expected treatment duration: 2-12 months
  Progress-scans once every 9 weeks will be performed
Description and change of Biomarker analysis/Pharmacodynamics | Day 1, 18, 25
  Blood biomarker analysis will be performed of PBMCs and where possible of tumor biposies performed during treatment
Pharmacogenetics | day 1 of treatment
  Full blood sample will be collected for pharmacogenetic analysis of important SNPs of drug disposition genes involved in the drug disposition of Nelfinivar and temsirolimus

CONTACTS AND LOCATIONS:
Overall Officials: Heinz-Josef Klumpen, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands